CLINICAL TRIAL: NCT01861756
Title: The Diabetes Medication Choice Cards Trial in Greece
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: European Foundation for the Study of Diabetes (Other); Mayo Clinic (Other)
Responsible Party: Principal Investigator, Apostolos Tsapas, Assistant Professor of Medicine, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AUTH87963; U1111-1138-2901 (Other: WHO - Universal Trial Number)
Record Dates: First submitted 2013-05-20; First posted 2013-05-24 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Shared Decision Making; Decision Aids
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (2):
- Diabetes Medication Choice Decision Aid (Experimental)
  Interventions: Other: Diabetes Medication Choice decision aid
- Standard care (No Intervention)

INTERVENTIONS:
Other: Diabetes Medication Choice decision aid — The Diabetes Medication Choice decision aid cards provide information about medications commonly used to treat type 2 diabetes mellitus. The tool was originally developed and successfully evaluated by Mayo Clinic researchers.
  Arms: Diabetes Medication Choice Decision Aid

SUMMARY:
A cluster randomized trial to assess the efficacy of the Diabetes Medication Choice decision aid among Greek patients with type 2 diabetes mellitus compared with usual care. The tool will serve as a facilitator for the Shared Decision Making process.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus for more than one year
* Agree to be followed for at least 6 months
* Willing to respond to survey questions immediately following the visit
* HbA1c value between 7.5% and 10%
* Need treatment intensification and there are more than one available treatment options

Exclusion Criteria:

* Decide not to intensify treatment or to intensify treatment through lifestyle modification, which is a sine qua non for diabetes treatment
* Is to transfer to another practice within the next 6 months
* Significant cognitive (e.g. dementia) or sensory limitations (e.g. blind) or other reasons (e.g. fatigue, limited attention, sleep deprivation) for which, in the judgment of the study personnel, they could not reasonably provide written informed consent or be able to use the decision aid
* Planning to enter a long-term care facility (e.g. nursing home) where medications will be administered by clinical personnel after hospital discharge
* Enrolled in other studies that require prolonged participation and follow-up
* Unable to speak Greek at a level necessary to complete the patient surveys and ensure involvement in decision making
* Women known to be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2013-05; Primary Completion 2014-02 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Apostolos Tsapas, MD, MSc, PhD, Principal Investigator — Aristotle University Of Thessaloniki
Locations (8):
- Greece (8):
  - Tzanio General Hospital, Piraeus, Attica
  - Private practice, Neapoli, Thessaloniki
  - Nea Michaniona Health Center, Néa Michanióna, Thessaloniki
  - Thermi S.A., Thermi, Thessaloniki
  - Alexandroupoli University Hospital, Alexandroupoli
  - NIMTS Military Hospital, Athens
  - Polikliniki General Hospital, Athens
  - Private practice, Serres

REFERENCES:
- [Derived] Karagiannis T, Liakos A, Branda ME, Athanasiadou E, Mainou M, Boura P, Goulis DG, LeBlanc A, Montori VM, Tsapas A. Use of the Diabetes Medication Choice Decision Aid in patients with type 2 diabetes in Greece: a cluster randomised trial. BMJ Open. 2016 Nov 14;6(11):e012185. doi: 10.1136/bmjopen-2016-012185. PMID 28186933

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diabetes Medication Choice Decision Aid | Usual Care
Started | 101 | 103
Completed | 88 | 85
Not Completed | 13 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diabetes Medication Choice Decision Aid | Usual Care | Total
Number analyzed (Participants) | 101 | 103 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (11) | 64.4 (11.3) | 65.1 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 61 | 116
  Male | 46 | 42 | 88
Region of Enrollment [Number; unit: participants]
  Greece | 101 | 103 | 204
Type 2 diabetes duration [Count of Participants; unit: Participants]
  <5 years | 27 | 22 | 49
  5 - 10 years | 20 | 27 | 47
  >10 years | 53 | 53 | 106
  missing data | 1 | 1 | 2
HbA1c [Mean (Standard Deviation); unit: %] | 8.4 (0.8) | 8.5 (0.8) | 8.5 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Overall Decisional Comfort (0-100, 100=no Conflict)
Description: Quality of the decision making process assessed by means of the Decisional Conflict Scale
Time Frame: Day 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Diabetes Medication Choice Decision Aid | Usual Care
Number analyzed (Participants) | 101 | 103
units on a scale | 82 [70 to 94] | 75.1 [61 to 89.2]

2. Secondary Outcome: Degree of Patient Knowledge About Available Treatment Alternatives
Description: Patients will complete a 6-item questionnaire addressing general knowledge about type 2 diabetes.
Time Frame: Day 1
Reporting Status: Not Posted

3. Secondary Outcome: Patient and Clinician Satisfaction With the Decision Making Process
Description: Patient satisfaction will be assessed using items from the Decisional Conflict Scale as well as two specific questions that require patients to assess the extent to which they would want for themselves and recommend to others similar decision support.
  Clinician satisfaction will be assessed using a 6-point likert-type question asking about their satisfaction regarding the discussion they had with their patient.
Time Frame: Day 1
Reporting Status: Not Posted

4. Secondary Outcome: Adherence With Antihyperglycemic Regimens as Reported by the Patient Himself/Herself or Assessed Utilizing the Pharmacy Records
Time Frame: 3 and 6 months after patient initial encounter
Reporting Status: Not Posted

5. Secondary Outcome: Glycemic Control (HbA1c)
Time Frame: 3 and 6 months after patient initial encounter
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Diabetes Medication Choice Decision Aid | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/103
Other Adverse Events (participants affected / at risk) | 0/101 | 0/103

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No